CLINICAL TRIAL: NCT00881803
Title: Implications of Concurrent Iron and Ascorbic Acid Supplementation on Iron Status in Persons With Spinal Cord Injury
Brief Title: Iron & Vitamin C Study
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: B4162C-6
Record Dates: First submitted 2009-03-25; First posted 2009-04-15 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injuries; Ascorbic Acid; Vitamin C; Iron; Dietary Supplements
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained for analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Ascorbic Acid Supplementation Only
- Group 2: Iron Supplementation Only
- Group 3: Concurrent Ascorbic Acid & Iron Supplementation

SUMMARY:
Iron overload is a life-threatening condition that can lead to liver disease, cardiac disease, diabetes and arthritis. Simultaneous supplementation with both iron and AA may place individuals with SCI at risk for iron overload as well as oxidative damage by iron-generated free radicals. Both conditions of high and low iron stores may present with common signs and symptoms. Accurate diagnosis of iron disorder should consider CRP, hematocrit, hemoglobin, serum iron, TIBC, percent saturation of iron binding capacity, serum ferritin and hepcidin.

The investigators are proposing a study to determine the effect of concurrent AA and iron supplementation on iron status of individuals with SCI. The investigators goal is to identify abnormal status that may be attributed to simultaneous supplementation of iron and AA to develop future supplementation protocols in this population for optimal iron status.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. 18 years to 90 years of age
3. Medically stable
4. Chronic SCI (>6 months post injury) without regard to the level or completeness of lesion
5. Supplementation with:

   * A standard recommended dose of 120-200 mg oral elemental iron (tablet or liquid; ferrous sulfate, fumarate or gluconate forms) for a minimum of 6 months; or
   * A standard recommended dose of 250-2,000 mg AA per day for a minimum of 6 months; or
   * Both 120-200 mg oral elemental iron AND 250-2,000 mg AA per day for a minimum of 6 months.
6. Veteran

Exclusion Criteria:

Acute cardiovascular, pulmonary or renal conditions

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: US Veterans with spinal cord injuries greater than 6 months who are located near Bronx, NY
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To determine iron status if supplemented with ascorbic acid (AA) and/or iron compared to supplementation with iron or AA. | 1 episode, at least 6 months after consistent ascorbic acid and/or iron supplementation

SECONDARY OUTCOMES:
Determine the prevalence of high iron status if receiving supplementation with both iron and AA compared to supplementation with iron or AA. | 1 episode, at least 6 months after consistent ascorbic acid and/or iron supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: William Bauman, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States